CLINICAL TRIAL: NCT02611817
Title: A Phase 3 Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Efficacy and Safety of Vedolizumab Subcutaneous as Maintenance Therapy in Subjects With Moderately to Severely Active Crohn's Disease Who Achieved Clinical Response Following Open-Label Vedolizumab Intravenous Therapy
Brief Title: Efficacy and Safety of Vedolizumab Subcutaneous (SC) as Maintenance Therapy in Crohn's Disease (CD)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MLN0002SC-3031; U1111-1168-0845 (Registry Identifier: WHO); 2015-000481-58 (EudraCT Number); NL55774.056.16 (Registry Identifier: CCMO); 16/LO/0090 (Registry Identifier: NRES); MLN0002SC-3031CTID (Registry Identifier: Israel); 163300410A0045 (Registry Identifier: NREC); 189748 (Registry Identifier: HC-CTD); MOH_2017-01-05_000039 (Other: CRS); JapicCTI-163386 (Registry Identifier: JapicCTI)
Record Dates: First submitted 2015-11-19; First posted 2015-11-23 (Estimated); Results first posted 2020-06-23 (Actual); Last update posted 2022-05-25 (Actual); Status verified 2022-05

CONDITIONS: Crohn's Disease
Keywords: Drug Therapy
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Vedolizumab SC 108 mg Maintenance Arm (Experimental): Open-label Induction: vedolizumab IV 300 milligram (mg), infusion at Week 0 (Day 1) and Week 2 (Day 15)
  Double-blind Maintenance: vedolizumab SC 108 mg injection once every 2 weeks (Q2W) starting at Week 6 up to Week 50
  Interventions: Drug: Vedolizumab SC 108 mg; Drug: Vedolizumab IV 300 mg
- Placebo SC Maintenance Arm (Placebo Comparator): Open-label Induction: vedolizumab IV 300 mg, infusion at Week 0 (Day 1) and Week 2 (Day 15)
  Double-blind Maintenance: matching placebo to vedolizumab SC injection Q2W starting at Week 6 up to Week 50
  Interventions: Drug: Placebo; Drug: Vedolizumab IV 300 mg

INTERVENTIONS:
Drug: Vedolizumab SC 108 mg — Vedolizumab SC Injection.
  Arms: Vedolizumab SC 108 mg Maintenance Arm
Drug: Placebo — Vedolizumab placebo-matching SC injection.
  Arms: Placebo SC Maintenance Arm
Drug: Vedolizumab IV 300 mg — Vedolizumab IV Injection.

SUMMARY:
The purpose of this study is to assess the effect of vedolizumab subcutaneous (vedolizumab SC) as maintenance treatment in participants with moderately to severely active CD who achieved clinical response following administration of vedolizumab intravenous (vedolizumab IV) induction therapy.

DETAILED DESCRIPTION:
The drug being tested in this study is called vedolizumab SC. Vedolizumab SC is being tested to treat people who have moderate to severely active CD. This study will look at clinical remission, as well as enhanced clinical response and corticosteroid-free remission in participants with CD who receive vedolizumab SC maintenance therapy after having achieved a clinical response to vedolizumab IV induction therapy.

The study will enroll approximately 824 participants. All participants will enter a 6 week Induction Phase where they will be administered open-label vedolizumab IV 300 mg via IV infusion at Week 0 (Day 1) and Week 2 (Day 15), and will then be assessed for a clinical response at Week 6. Participants who achieve a clinical response at Week 6 will be randomly assigned to one of the two treatment groups:

* Vedolizumab SC 108 mg Maintenance Arm
* Placebo SC Maintenance Arm

Participants who do not achieve a clinical response will not be randomized into the Maintenance Period, and instead will receive a third infusion of vedolizumab IV 300 mg at Week 6.

This multi-center trial will be conducted worldwide. The overall time to participate in this study is up to 71 weeks. Participants will make multiple visits to the clinic, plus a final visit 18 weeks after last dose of study drug for a follow-up assessment. Participants will also participate in a long-term safety follow-up, by phone, at 6 months after the last dose of study drug.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of CD established at least 3 months prior to screening by clinical and endoscopic evidence corroborated by a histopathology report.
2. Moderately to severely active CD as determined by a CDAI score of 220 to 450 and 1 of the following:

   * C-reactive protein (CRP) level greater than (>) 2.87 milligram per liter (mg/L) OR
   * Ileocolonoscopy with photographic documentation of a minimum of 3 nonanastomotic ulcerations (each >0.5 centimeter [cm] in diameter) or 10 aphthous ulcerations (involving a minimum of 10 contiguous cm of intestine) consistent with CD OR
   * Fecal calprotectin >250 microgram per gram (mcg/g) stool during the screening period in conjunction with computed tomography enterography (CTE), magnetic resonance enterography (MRE), contrast-enhanced small bowel radiography, or wireless capsule endoscopy revealing CD ulcerations (aphthae not sufficient).
3. CD involvement of the ileum and/or colon, at a minimum.
4. Inadequate response with, loss of response to, or intolerance to corticosteroids, immunomodulators, or Tumor necrosis factor-alpha (TNF-α) antagonists.

Exclusion Criteria:

1. Evidence of abdominal abscess at Screening.
2. Extensive colonic resection, subtotal or total colectomy.
3. History of >3 small bowel resections or diagnosis of short bowel syndrome.
4. Ileostomy, colostomy, or known fixed symptomatic stenosis of the intestine.
5. Prior exposure to investigational or approved non-biologic therapies (example, cyclosporine, tacrolimus, thalidomide, or tofacitinib) for the treatment of underlying disease within 30 days or 5 half-lives of screening (whichever is longer).
6. Prior exposure to any investigational or approved biologic or biosimilar agent within 60 days or 5 half-lives of screening (whichever is longer).
7. Prior exposure to vedolizumab.
8. Surgical intervention for CD required at any time during the study.
9. History or evidence of adenomatous colonic polyps that have not been removed, or of colonic mucosal dysplasia.
10. Suspected or confirmed diagnosis of ulcerative colitis, indeterminate colitis, ischaemic colitis, radiation colitis, diverticular disease associated with colitis, or microscopic colitis.
11. Active infections.
12. Chronic hepatitis B virus (HBV) or C (HCV) infection, tuberculosis (TB) (active or latent), or congenital or acquired immunodeficiency. HBV immune participants (that is, being hepatitis B surface antigen [HBsAg] negative and hepatitis B antibody positive) may, however, be included.
13. History of any major neurological disorders, including stroke, multiple sclerosis, brain tumor, or neurodegenerative disease.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 644 (Actual)
Dates: Start 2016-01-04 (Actual); Primary Completion 2019-05-06 (Actual); Study Completion 2019-08-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director Clinical Science, Study Director — Takeda
Locations (194):
- United States (30):
  - Arizona Arthritis & Rheumatology Research, PLLC, Phoenix, Arizona
  - Medical Research Center of Connecticut, LLC, Hamden, Connecticut
  - Middlesex Gastroenterology Associates, Middletown, Connecticut
  - Nature Coast Clinical Research, LLC, Inverness, Florida
  - L & L Research Choices, Inc., Miami, Florida
  - Gastroenterology Group of Naples, Naples, Florida
  - Shafran Gastroenterology Center, Winter Park, Florida
  - Atlanta Gastroenterology Associates, Atlanta, Georgia
  - Gastroenterology Associates of Central Georgia, Macon, Georgia
  - Atlanta Gastroenterology Specialists, PC, Suwanee, Georgia
  - Grand Teton Research Group, PLL, Idaho Falls, Idaho
  - Rush University Medical Center, Chicago, Illinois
  - Carle Foundation Hospital, Urbana, Illinois
  - Cotton-O'Neil Clinical Research Center, Digestive Health, Topeka, Kansas
  - Tri-State Gastroenterology Associates, Crestview Hills, Kentucky
  - Gastroenterology Associates, LLC, Baton Rouge, Louisiana
  - Louisiana Research Center, LLC, Shreveport, Louisiana
  - Metropolitan Gastroenterology Group, PC, Chevy Chase Clinical Research, Chevy Chase, Maryland
  - Clinical Research Institute of Michigan, LLC, Chesterfield, Michigan
  - Gastroenterology Associates of Western Michigan, P.L.C., Wyoming, Michigan
  - Mayo Clinic - Rochester, Rochester, Minnesota
  - Ehrhardt Clinical Research, LLC, Belton, Missouri
  - Long Island Clinical Research Associates, Great Neck, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Gastro-Enterology Research of Lima, Lima, Ohio
  - Options Health Research, Tulsa, Oklahoma
  - Gastroenterology Center of the MidSouth PC, Germantown, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - San Antonio Gastroenterology, San Antonio, Texas
  - Allegiance Research Specialists, LLC, Milwaukee, Wisconsin
- Australia (9):
  - Concord Repatriation General Hospital, Concord, New South Wales
  - Nepean Hospital, Kingswood, New South Wales
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Tennyson Centre Day Hospital, Bedford Park, South Australia
  - Ballarat Base Hospital, Ballarat, Victoria
  - Royal Melbourne Hospital, Melbourne, Victoria
  - The Alfred Hospital, Melbourne, Victoria
  - Fiona Stanley Hospital, Murdoch, Western Australia
  - St John of God Subiaco Hospital, Subiaco, Western Australia
- Belgium (5):
  - Imeldaziekenhuis, Bonheiden
  - Universitair Ziekenhuis Gent, Ghent
  - AZ Groeninge - Kennedylaan, Kortrijk
  - ZNA Jan Palfijn, Merksem
  - AZ Delta, Roeselare
- Bosnia and Herzegovina (2):
  - University Clinical Centre of the Republic of Srpska, Banja Luka
  - University Clinical Hospital Mostar, Mostar
- Brazil (8):
  - Instituto Goiano de Gastroenterologia e Endoscopia Digestiva Ltda, Goiânia, Goiás
  - HUGG - Hospital Universitario Gaffree e Guinle, Rio de Janeiro, Rio Do Janeiro
  - HUCFF-UFRJ - Hospital Universitario Clementino Fraga Filho - Universidade Federal do Rio de Janeiro, Rio de Janeiro, Rio Do Janeiro
  - Hospital de Clinicas de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - UNESP - Faculdade de Medicina da Universidade Estadual Paulista - Campus Botucatu, Botucatu, São Paulo
  - Faculdade de Medicina do ABC, Santo André, São Paulo
  - Irmandade da Santa Casa da Misericordia de Santos, Santos, São Paulo
  - Fundacao Faculdade Regional de Medicina de Sao Jose do Rio Preto, São José do Rio Preto, São Paulo
- Bulgaria (5):
  - MHAT "Hadzhi Dimitar", OOD, Sliven
  - "City Clinic UMHAC" EOOD, Sofia
  - UMHAT "Sv. Ivan Rilski", EAD, Sofia
  - UMHAT 'Tsaritsa Yoanna - ISUL', EAD, Sofia
  - Fourth MHAT - Sofia EAD, Sofia
- Canada (5):
  - Zeidler Ledcor Centre - University of Alberta, Edmonton, Alberta
  - PerCuro Clinical Research Ltd., Victoria, British Columbia
  - LHSC - University Hospital, London, Ontario
  - LHSC - Victoria Hospital, London, Ontario
  - Toronto Digestive Disease Associates, Inc., Vaughan, Ontario
- Czechia (5):
  - CCBR - Czech Brno, s.r.o.., Brno
  - Hepato-Gastroenterologie HK s.r.o., Hradec Králové
  - A-SHINE s.r.o., Pilsen
  - CCBR Czech Prague, s.r.o., Prague
  - Axon Clinical s.r.o., Prague
- Denmark (2):
  - Odense Universitetshospital, Odense C
  - Regionshospitalet Silkeborg, Silkeborg
- North Estonia Medical Centre Foundation, Tallinn, Estonia
- Germany (5):
  - Medizinische Hochschule Hannover, Hanover, Lower Saxony
  - Universitaetsmedizin der Johannes Gutenberg-Universitaet Mainz, Mainz, Rhineland-Palatinate
  - EUGASTRO GmbH, Leipzig, Saxony
  - DRK Kliniken Berlin Westend, Berlin
  - Krankenhaus Waldfriede e. V., Berlin
- Hungary (9):
  - Obudai Egeszsegugyi Centrum Kft., Budapest
  - Semmelweis Egyetem, Budapest
  - Szent Janos Korhaz es Eszak-budai Egyesitett Korhazak, Budapest
  - Pannonia Maganorvosi Centrum, Budapest
  - Pest Megyei Flor Ferenc Korhaz, Kistarcsa
  - Borsod-Abauj-Zemplen Megyei Kozponti Korhaz es Egyetemi Oktatokorhaz, Miskolc
  - Karolina Korhaz-Rendelointezet, Mosonmagyaróvár
  - Tolna Megyei Balassa Janos Korhaz, Szekszárd
  - Fejer Megyei Szent Gyorgy Egyetemi Oktato Korhaz, Székesfehérvár
- Israel (6):
  - HaEmek Medical Center, Afula
  - Soroka University Medical Center, Beersheba
  - Shaare Zedek Medical Center, Jerusalem
  - Chaim Sheba Medical Center, Ramat Gan
  - Kaplan Medical Center, Rehovot
  - Tel Aviv Sourasky Medical Center, Tel Aviv
- Italy (10):
  - IRCCS Ospedale Casa Sollievo della Sofferenza, San Giovanni Rotondo, Foggia
  - I.R.C.C.S Policlinico San Donato, San Donato Milanese (MI), Milano
  - Azienda Ospedaliera Universitaria Policlinico Sant'Orsola Malpighi, Bologna
  - Azienda Ospedaliera Ospedale Cannizzaro, Catania
  - Azienda Socio Sanitaria Territoriale Fatebenefratelli (Presidio Ospedale Sacco), Milan
  - A.O.U. Policlinico di Modena, Modena
  - Azienda Ospedaliera di Padova, Padua
  - Azienda Ospedaliera Vincenzo Cervello, Palermo
  - Azienda Ospedaliera San Camillo Forlanini, Roma
  - Policlinico Universitario Agostino Gemelli, Roma
- Japan (14):
  - Toho University Sakura Medical Center, Sakura-shi, Chiba
  - Fukuoka University Chikushi Hospital, Chikushino-shi, Fukuoka
  - Tokushukai Sapporo Tokushukai Hospital, Sapporo, Hokkaido
  - Sapporo-Kosei General Hospital, Sapporo, Hokkaido
  - Tokushukai Sapporo Higashi Tokushukai Hospital, Sapporo, Hokkaido
  - Hyogo College of Medicine Hospital, Nishinomiya-shi, Hyōgo
  - Iwate Medical University Hospital, Morioka, Iwate
  - Gokeikai Ofuna Chuo Hospital, Kamakura-shi, Kanagawa
  - Kinshukai Infusion Clinic, Osaka, Osaka
  - Saga University Hospital, Saga, Saga-ken
  - Hamamatsu South Hospital, Hamamatsu, Shizuoka
  - Kitasato University Kitasato Institute Hospital, Minatoku, Tokyo-To
  - JCHO Tokyo Yamate Medical Center, Shinjuku-ku, Tokyo-To
  - Wakayama Medical University Hospital, Wakayama, Wakayama
- Lithuania (2):
  - Hospital of Lithuanian University of Health Sciences Kaunas Clinics, Kaunas
  - Vilnius University Hospital Santariskiu Clinic, Public Institution, Vilnius
- Mexico (4):
  - Morales Vargas Centro de Investigacion, S.C., León, Guanajuato
  - Centro de Investigacion Farmacologica del Bajio, S.C., León, Guanajuato
  - Instituto de Investigaciones Aplicadas a la Neurociencia A.C., Durango
  - Sociedad de Metabolismo y Corazon S.C, Veracruz
- Netherlands (3):
  - Academisch Medisch Centrum, Amsterdam
  - Albert Schweitzer Ziekenhuis, Dordwijk, Dordrecht
  - Erasmus Medisch Centrum, Rotterdam
- Poland (12):
  - NZOZ Vitamed, Bydgoszcz
  - Gabinet Endoskopii Przewodu Pokarmowego, Krakow
  - SPZOZ Uniwersytecki Szpital Klin. nr 1 im.N.Barlickiego UM, Lodz
  - Santa Familia Centrum Badan, Profilaktyki i Leczenia, Lodz
  - GASTROMED Sp. z o.o., Lublin
  - Twoja Przychodnia-Szczecinskie Centrum Medyczne, Szczecin
  - Centrum Zdrowia MDM, Warsaw
  - Centralny Szpital Kliniczny MSW w Warszawie, Warsaw
  - Centrum Onkologii-Instytut im. M. Sklodowskiej Curie, Warsaw
  - Nzoz Vivamed, Warsaw
  - LexMedica Osrodek Badan Klinicznych, Wroclaw
  - Ars-Medica S.C Rybak Maria, Rybak Zbigniew, Wroclaw
- Romania (3):
  - Spitalul Clinic Colentina, Bucharest
  - Institutul Clinic Fundeni, Bucharest
  - S.C Centrul de Gastroenterologie Dr. Goldis S.R.L, Timișoara
- Russia (11):
  - Kazan State Medical University, Kazan'
  - TSBIH "Territorial Clinical Hospital", Krasnoyarsk
  - SBEIHPE Novosibirsk State Medical University, Novosibirsk
  - FSBSI "Scientific and Research Institute of Physiology and Basic Medicine", Novosibirsk
  - BHI of Omsk region Clinical Oncology Dispensary, Omsk
  - SBEI of HPE "Omsk SMA" SBEI HPE "Omsk State Medical University" of the MoH of the RF, Omsk
  - SBEI HPE "Rostov State Medical University" of the MoH of the RF, Rostov-on-Don
  - SPb SBIH "City Hospital of Saint Martyr Elizaveta", Saint Petersburg
  - LLC "RIAT SPb", Saint Petersburg
  - SPb SBIH "City Hospital # 40 of Kurortnyi region", Sestroretsk
  - SBIH of Yaroslavl region " Regional Clinical Hospital ", Yaroslavl
- Serbia (5):
  - Clinical Helth Centre Zvezdara, Belgrade
  - Military Medical Academy, Belgrade
  - Clinical Center Bezanijska kosa, Belgrade
  - Clinical Center Kragujevac, Kragujevac
  - Clinical Center of Vojvodina, Novi Sad
- Slovakia (2):
  - Fakultna nemocnica s poliklinikou F.D. Roosevelta, Banská Bystrica
  - Univerzitna nemocnica Bratislava, Nemocnica Ruzinov, Bratislava
- South Africa (2):
  - Dr CCM Ziady Practice, Pretoria, Gauteng
  - Dr JP Wright Practice, Cape Town, Western Cape
- South Korea (8):
  - Kyungpook National University Hospital, Daegu
  - Yeungnam University Hospital, Daegu
  - Kyung Hee University Hospital, Seoul
  - Seoul National University Hospital, Seoul
  - Kangbuk Samsung Hospital, Seoul
  - Severance Hospital, Yonsei University, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
- Karolinska Universitetssjukhuset - Solna, Stockholm, Sweden
- Mackay Memorial Hospital, Taipei, Taiwan
- Turkey (Türkiye) (5):
  - Ankara University Medical Faculty, Ankara
  - Haydarpasa Numune Training and Research Hospital, Istanbul
  - Marmara University Pendik Research and Training Hospital, Istanbul
  - Kocaeli Derince Training and Research Hospital, Kocaeli
  - Mersin University Medical Faculty, Mersin
- Ukraine (14):
  - RCI Chernivtsi RCH Dep of Surgery HSEI of Ukr Bukovinian SMU, Chernivtsi
  - SI Institute of Gastroenterology of NAMSU Dept of Stomach & Duodenum Diseases, D&ThN SI DMA of MoHU, Dnipro
  - CNE Prof. O.O. Shalimov Kharkiv City Clinical Hospital #2 of KCC, Kharkiv
  - CI A.and O. Tropiny City Clinical Hospital, Kherson
  - Kyiv CCH #12 Dept of Therapy O.O.Bogomolets NMU, Kyiv
  - CI of Kyiv RC Kyiv Regional Clinical Hospital, Kyiv
  - MI of Healthcare Kyiv RCH P.L. Shupyk NMA of PGE, Kyiv
  - Communal City Clinical Hospital of Ambulance, Dept of Therapy #1 D.Halytskyi Lviv NMU, Lviv
  - CI Odesa Regional Clinical Hospital, Odesa
  - Ternopil University Hospital, Ternopil
  - Private Small Enterprise Medical Center Pulse, Vinnytsia
  - Vinnytsia RCH of Veterans of War Dept of Therapy#1 Vinnytsia M.I.Pyrogov NMU, Vinnytsia
  - MCIC MC LLC Health Clinic, Vinnytsia
  - CI City Hospital #1, Zaporizhzhia
- United Kingdom (5):
  - Royal Devon and Exeter Hospital (Wonford), Exeter, Devon
  - St George's Hospital, London, Greater London
  - Whipps Cross University Hospital, London, Greater London
  - Royal Shrewsbury Hospital, Shrewsbury, Shropshire
  - University Hospital Coventry, Coventry, West Midlands

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/ For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- [Derived] D'Haens G, Baert F, Danese S, Kobayashi T, Loftus EV Jr, Sandborn WJ, Dornic Q, Lindner D, Kisfalvi K, Marins EG, Vermeire S. Efficacy of vedolizumab during intravenous induction therapy in ulcerative colitis and Crohn's disease: post hoc analysis of patient-reported outcomes from the VISIBLE 1 and 2 studies. Eur J Gastroenterol Hepatol. 2024 Apr 1;36(4):404-415. doi: 10.1097/MEG.0000000000002728. Epub 2024 Feb 21. PMID 38417060

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with moderate to severe Crohn's disease (CD) took part in the study at 169 investigative sites in North America, South America, Western/Northern Europe, Central Europe, Eastern Europe, East Asia, and Africa/Australia from 04 Jan 2016 to 06 Aug 2019.
Pre-assignment Details: Participants were enrolled in open-label (OL) induction phase to receive vedolizumab (VDZ) intravenous (IV). Participants with clinical response (CR) at Week 6 were randomized into double-blind maintenance phase to receive VDZ subcutaneous/placebo, and who did not achieve CR at Week 6 received 3rd infusion of OL VDZ IV and completed Week 14 visit.
Groups:
- Open-label Induction Phase: Vedolizumab 300 mg IV: Vedolizumab 300 milligram (mg), infusion, intravenously, once at Weeks 0, 2 in the open-label induction phase.
- Maintenance Phase: Induction IV + Placebo: Vedolizumab placebo-matching injection, subcutaneously, once every 2 weeks from Week 6 up to Week 50. Participants who received vedolizumab 300 mg IV infusion in open-label induction phase and achieved clinical response at Week 6 were randomized to receive placebo in maintenance phase.
- Maintenance Phase: Induction IV + Vedolizumab 108 mg SC: Vedolizumab 108 mg, injection, subcutaneously, once every 2 weeks from Week 6 up to Week 50. Participants who received vedolizumab 300 mg IV infusion in open-label induction phase and achieved clinical response at Week 6 were randomized to receive vedolizumab injection subcutaneously in maintenance phase.
Period: Open-label Induction Phase
Arm/Group | Open-label Induction Phase: Vedolizumab 300 mg IV | Maintenance Phase: Induction IV + Placebo | Maintenance Phase: Induction IV + Vedolizumab 108 mg SC
Started | 644 | 0 | 0
Completed (Completers included participants who received OL vedolizumab IV and had Week 14 visit.) | 594 | 0 | 0
Not Completed | 50 | 0 | 0
Not completed — Reason not Specified | 9 | 0 | 0
Not completed — Lack of Efficacy | 8 | 0 | 0
Not completed — Pregnancy | 1 | 0 | 0
Not completed — Withdrawal by Subject | 9 | 0 | 0
Not completed — Lost to Follow-up | 2 | 0 | 0
Not completed — Protocol Violation | 5 | 0 | 0
Not completed — Adverse Event | 16 | 0 | 0
Period: Double-blind Maintenance Phase
Arm/Group | Open-label Induction Phase: Vedolizumab 300 mg IV | Maintenance Phase: Induction IV + Placebo | Maintenance Phase: Induction IV + Vedolizumab 108 mg SC
Started (Participants who achieved clinical response at Week 6 entered the Maintenance Phase.) | 0 | 135 | 275
Completed | 0 | 73 | 168
Not Completed | 0 | 62 | 107
Not completed — Adverse Event | 0 | 12 | 11
Not completed — Randomized but not Treated | 0 | 1 | 0
Not completed — Reason not Specified | 0 | 1 | 2
Not completed — Lack of Efficacy | 0 | 43 | 78
Not completed — Pregnancy | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 5 | 14
Not completed — Lost to Follow-up | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: The safety analysis set-combined (SAF-C) included all participants who received at least 1 dose of study vedolizumab IV.
Groups:
- Induction Phase Only: Vedolizumab 300 mg IV: Vedolizumab 300 mg, infusion, intravenously, once at Weeks 0, 2 in the open-label induction phase Participants who did not achieve clinical response at Week 6 received third infusion of vedolizumab 300 mg IV on Week 6.
- Total: Total of all reporting groups
Arm/Group | Induction Phase Only: Vedolizumab 300 mg IV | Maintenance Phase: Induction IV + Placebo | Maintenance Phase: Induction IV + Vedolizumab 108 mg SC | Total
Number analyzed (Participants) | 235 | 134 | 275 | 644
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.4 (12.79) | 36.1 (12.93) | 38.2 (13.85) | 37.5 (13.29)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 119 | 68 | 118 | 305
  Male | 116 | 66 | 157 | 339
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 2 | 3
  Not Hispanic or Latino | 50 | 20 | 60 | 130
  Unknown or Not Reported | 185 | 113 | 213 | 511
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 2 | 0 | 2
  Asian | 23 | 6 | 17 | 46
  Native Hawaiian or Other Pacific Islander | 2 | 1 | 0 | 3
  Black or African American | 3 | 1 | 7 | 11
  White | 207 | 124 | 250 | 581
  More than one race | 0 | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0
Weight [Mean (Standard Deviation); unit: kilogram (kg)] | 69.94 (18.403) | 69.79 (18.103) | 74.08 (18.994) | 71.68 (18.684)
Body Mass Index [Mean (Standard Deviation); unit: kilogram per square meter (kg/m^2)] | 24.20 (6.073) | 23.93 (5.541) | 25.06 (5.915) | 24.51 (5.909)
Smoking Classification [Count of Participants; unit: Participants]
  Never smoked | 140 | 85 | 148 | 373
  Current smoker | 49 | 26 | 54 | 129
  Ex-smoker | 46 | 23 | 73 | 142

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving Clinical Remission at Week 52
Description: Clinical remission is defined as a Crohn's Disease Activity Index (CDAI) score less than or equal to (<=) 150 at Week 52. A CDAI is a multi-item instrument which measures severity of active Crohn's Disease monitored over 7 days includes participant reported symptoms, physician-assessed signs, and laboratory markers. CDAI score is equal to (=) sum of weighted scores for subjective items (number of liquid/soft stools, degree of abdominal pain, general well-being); and objective items (use of anti-diarrhoeal medication, abdominal mass, haematocrit, presence of extraintestinal manifestation, body weight). CDAI scores range approximately from 0 to 600, higher scores indicating greater disease activity.
Time Frame: Week 52
Population: The full analysis set (FAS): All randomized participants who received at least 1 dose of study SC drug (placebo or VDZ). Participants who only received induction IV therapy and were not randomized into the maintenance phase were not included in FAS. Participants in this set were analyzed according to the treatment they were randomized to receive.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Maintenance Phase: Induction IV + Placebo | Maintenance Phase: Induction IV + Vedolizumab 108 mg SC
Number analyzed (Participants) | 134 | 275
percentage of participants | 34.3 [26.3 to 43.0] | 48.0 [42.0 to 54.1]
Statistical Analysis 1: Comparison: Maintenance Phase: Induction IV + Placebo vs Maintenance Phase: Induction IV + Vedolizumab 108 mg SC; P-value was calculated by Cochran-Mantel-Haenszel (CMH) test stratified by electronic data capture (EDC) stratum according to concomitant use of corticosteroids, clinical remission status at Week 6, and previous TNF-alpha antagonist failure/exposed or concomitant immunomodulator use; Test type: Superiority; p = 0.008, Cochran-Mantel-Haenszel; Clopper-Pearson method = 13.7, 95% CI 2-sided [3.8 to 23.7]

2. Secondary Outcome: Percentage of Participants Achieving Enhanced Clinical Response at Week 52
Description: Enhanced clinical response is defined as a decrease from Baseline of greater than or equal to (>=) 100 points in the CDAI score at Week 52. A CDAI is a multi-item instrument which measures severity of active CD monitored over 7 days includes participant reported symptoms, physician-assessed signs, and laboratory markers. CDAI score = Sum of weighted scores for subjective items (number of liquid/soft stools, degree of abdominal pain, general well-being); and objective items (use of anti-diarrhoeal medication, abdominal mass, haematocrit, presence of extraintestinal manifestation, body weight). CDAI scores range approximately from 0 to 600, higher scores indicating greater disease activity.
Time Frame: Week 52
Population: The FAS included all randomized participants who received at least 1 dose of study SC drug (placebo or VDZ). Participants who only received induction IV therapy and were not randomized into the maintenance phase were not included in FAS. Participants in this set were analyzed according to the treatment they were randomized to receive.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Maintenance Phase: Induction IV + Placebo | Maintenance Phase: Induction IV + Vedolizumab 108 mg SC
Number analyzed (Participants) | 134 | 275
percentage of participants | 44.8 [36.2 to 53.6] | 52.0 [45.9 to 58.0]
Statistical Analysis 1: Comparison: Maintenance Phase: Induction IV + Placebo vs Maintenance Phase: Induction IV + Vedolizumab 108 mg SC; P-value was calculated by CMH test stratified by EDC stratum according to concomitant use of corticosteroids, clinical remission status at Week 6, and previous TNF-alpha antagonist failure/exposed or concomitant immunomodulator use; Test type: Superiority; p = 0.167, Cochran-Mantel-Haenszel; Clopper-Pearson method = 7.3, 95% CI 2-sided [-3.0 to 17.5]

3. Secondary Outcome: Percentage of Participants Achieving Corticosteroid-free Remission at Week 52
Description: Corticosteroid-free remission is defined as participants using oral corticosteroids at Baseline (Week 0) who have discontinued oral corticosteroids and are in clinical remission at Week 52. Clinical remission is defined as a CDAI score <=150 at Week 52. CDAI score = Sum of weighted scores for subjective items (number of liquid/soft stools, degree of abdominal pain, general well-being); and objective items (use of anti-diarrhoeal medication, abdominal mass, haematocrit, presence of extraintestinal manifestation, body weight). CDAI scores range approximately from 0 to 600, higher scores indicating greater disease activity.
Time Frame: Week 52
Population: Participants from FAS, who used concomitant oral corticosteroid at Baseline. FAS had all participants who received at least 1 dose of SC drug. Participants who only received induction IV therapy and were not randomized into maintenance phase were not included in FAS. Participants were analyzed according to randomized treatment assignment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Maintenance Phase: Induction IV + Placebo | Maintenance Phase: Induction IV + Vedolizumab 108 mg SC
Number analyzed (Participants) | 44 | 95
percentage of participants | 18.2 [8.2 to 32.7] | 45.3 [35.0 to 55.8]
Statistical Analysis 1: Comparison: Maintenance Phase: Induction IV + Placebo vs Maintenance Phase: Induction IV + Vedolizumab 108 mg SC; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.002, Cochran-Mantel-Haenszel; Clopper-Pearson method = 27.1, 95% CI 2-sided [11.9 to 42.3]

4. Secondary Outcome: Percentage of TNF-alpha Antagonist Naive Participants Achieving Clinical Remission at Week 52
Description: Clinical remission is defined as CDAI score <=150 at Week 52. CDAI score = Sum of weighted scores for subjective items (number of liquid/soft stools, degree of abdominal pain, general well-being); and objective items (use of anti-diarrhoeal medication, abdominal mass, haematocrit, presence of extraintestinal manifestation, body weight). CDAI scores range approximately from 0 to 600, higher scores indicating greater disease activity.
Time Frame: Week 52
Population: Participants from FAS, who were TNF-alpha antagonist naïve and had clinical remission. FAS had all participants who received at least 1 dose of SC drug. Participants who only received induction IV therapy and were not randomized in maintenance phase were not included in FAS. Participants were analyzed according to randomized treatment assignment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Maintenance Phase: Induction IV + Placebo | Maintenance Phase: Induction IV + Vedolizumab 108 mg SC
Number analyzed (Participants) | 63 | 107
percentage of participants | 42.9 [30.5 to 56.0] | 48.6 [38.8 to 58.5]
Statistical Analysis 1: Comparison: Maintenance Phase: Induction IV + Placebo vs Maintenance Phase: Induction IV + Vedolizumab 108 mg SC; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.591, Cochran-Mantel-Haenszel; Clopper-Pearson method = 4.3, 95% CI 2-sided [-11.6 to 20.3]

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events are adverse events that started after the first dose of study drug up to 18 weeks after the last dose of study drug (up to Week 68)
Description: At each visit investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant/observed by the investigator was recorded, irrespective of the relation to study treatment. Participants were regrouped to mirror the baseline groupings for the better readability of the complex design. All participants and events (collected during the study in the induction/maintenance phase) have been accounted for the groupings.
Arm/Group | Induction Phase Only: Vedolizumab 300 mg IV | Maintenance Phase: Induction IV + Placebo | Maintenance Phase: Induction IV + Vedolizumab 108 mg SC
All-Cause Mortality (participants affected / at risk) | 0/235 | 0/134 | 0/275
Serious Adverse Events (participants affected / at risk) | 39/235 | 14/134 | 23/275
Other Adverse Events (participants affected / at risk) | 40/235 | 54/134 | 102/275
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Induction Phase Only: Vedolizumab 300 mg IV (N=235) | Maintenance Phase: Induction IV + Placebo (N=134) | Maintenance Phase: Induction IV + Vedolizumab 108 mg SC (N=275)
Anaemias (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 1 (2)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Angina pectoris (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Crohn's disease (Gastrointestinal disorders) | 14 (14) | 5 (7) | 6 (7)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 2 (3) | 1 (1)
Ileal stenosis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Anal fistula (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1)
Enterovesical fistula (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2)
Subileus (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
General physical health deterioration (General disorders) | 0 (0) | 0 (0) | 1 (1)
Anal abscess (Infections and infestations) | 2 (2) | 1 (1) | 1 (1)
Abdominal wall abscess (Infections and infestations) | 1 (1) | 1 (2) | 0 (0)
Abscess intestinal (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Rectal abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Dengue fever (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Gastrointestinal anastomotic complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Incisional hernia (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
White blood cell count increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Weight gain poor (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Intraductal papilloma of breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Haemorrhagic stroke (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Intraventricular haemorrhage (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Alcoholism (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Enterocutaneous fistula (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0)
Jejunal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Large intestinal ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Large intestine perforation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal abscess (Infections and infestations) | 4 (6) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Colonic abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Perirectal abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Hepatitis cholestatic (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Hemiparesis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Hemiplegia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal anastomotic stenosis (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Ureterolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Induction Phase Only: Vedolizumab 300 mg IV (N=235) | Maintenance Phase: Induction IV + Placebo (N=134) | Maintenance Phase: Induction IV + Vedolizumab 108 mg SC (N=275)
Crohn's disease (Gastrointestinal disorders) | 7 (7) | 23 (25) | 36 (36)
Abdominal pain (Gastrointestinal disorders) | 9 (11) | 11 (14) | 21 (25)
Nausea (Gastrointestinal disorders) | 9 (10) | 7 (7) | 11 (14)
Vomiting (Gastrointestinal disorders) | 4 (5) | 7 (8) | 6 (7)
Nasopharyngitis (Infections and infestations) | 7 (8) | 6 (8) | 25 (26)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 5 (6) | 17 (23)
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 (8) | 9 (10) | 17 (21)
Headache (Nervous system disorders) | 10 (10) | 5 (9) | 15 (19)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.

DOCUMENTS (2):
  • Study Protocol (2017-08-24): https://cdn.clinicaltrials.gov/large-docs/17/NCT02611817/Prot_000.pdf
  • Statistical Analysis Plan (2019-06-24): https://cdn.clinicaltrials.gov/large-docs/17/NCT02611817/SAP_001.pdf